CLINICAL TRIAL: NCT02309983
Title: Activity Dependent Rehabilitation Model In Incomplete Spinal Cord Injury: Neuromuscular and Skeletal Changes
Brief Title: Activity Dependent Rehabilitation Model to Improve Bone and Muscle Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Gail Forrest, Assistant Director Human Performance Engineering Lab, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-3063-SCR-E-0
Record Dates: First submitted 2013-09-05; First posted 2014-12-05 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Disuse Osteoporosis; Atrophy, Disuse; Nervous System; Structural; Marker; Skeletal Muscle Hypertrophy
Keywords: bone turnover; muscle atrophy; fiber
MeSH Terms: conditions — Muscular Disorders, Atrophic; Neurologic Manifestations; Muscular Atrophy | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electrical Stimulation Alone Group (Active Comparator): Group 1 will receive 1hr of electrical stimulation while lying down followed by 15 min of overground training. Electrical stimulation will be applied through leads and self-adhesive electrodes over muscles of both legs. Two electrodes will be used for each muscle. Electrical stimulation will be induced by using the EMPI, Inc., St. Paul, MN [Respond Select Neuromuscular Stimulation]. There will be 60 sessions/3x week for 20 weeks.
  Interventions: Other: Electrical Stimulation
- Stand Retraining Alone with BWS (Placebo Comparator): Group 2 will receive standing retraining with BWS alone on a treadmill without functional electrical stimulation. Locomotor training consists of (step training and stand retraining) on the treadmill, over ground training, and community ambulation. BWS will be given when a subject can not maintain his/her body weight while executing limb locomotion. BWS will be given when a subject can not maintain his/her body weight while executing limb locomotion. The duration of stand retraining sessions will be up to 1 hour or determined by subject's fatigue. There will be 60 sessions/3x week for 20 weeks.
  Interventions: Other: Stand Retraining with Body Weight Support (BWS)
- Stand Retraining and ES Group (Experimental): Group 3 will receive standing retraining with BWS with electrical stimulation, followed by 15 min of overground training. Locomotor training consists of (step training and stand retraining) on the treadmill, over ground training, and community ambulation. BWS will be given when a subject can not maintain his/her body weight while executing limb locomotion. Electrical stimulation will start while participant is seated and before he/she is brought up to full standing. There will be 60 sessions/3x week for 20 weeks.
  Interventions: Other: Electrical Stimulation; Other: Stand Retraining with Body Weight Support (BWS)

INTERVENTIONS:
Other: Electrical Stimulation — Electrical stimulation is a rehabilitative approach that generates muscle activity by alternating leg extension and flexion even in individuals who are unable to stand or step independently. Electrical stimulation will be applied to multiple muscles of the lower limb.
  Arms: Electrical Stimulation Alone Group; Stand Retraining and ES Group
Other: Stand Retraining with Body Weight Support (BWS) — Locomotor training consists of (step training and stand retraining) on the treadmill, over ground training, and community ambulation. BWS will be given when a subject can not maintain his/her body weight while executing limb locomotion.
  Other Names: Locomotor Training
  Arms: Stand Retraining Alone with BWS; Stand Retraining and ES Group

SUMMARY:
For many after spinal cord injury (SCI) there is immobilization, muscle atrophy, bone loss, fracture risk during transferring (or falls), and the risk of secondary complications, and increase in attendance care and cost. It is important to develop multi dimensional rehabilitation strategies for people after SCI to enhance functional recovery towards walking, and enhance an increase in muscle and bone to potentially prepare the injured nervous system in the event of a cure. Locomotor training (Stand retraining and step re training) an activity-based rehabilitative approach generates muscle activity and provides weight bearing and joint contact kinetics, even in individuals who are unable to stand or step independently. Cross-sectional animal and human SCI studies have demonstrated that locomotor training (LT) (stand retraining and step retraining using body weight support treadmill training) has improved the capacity to stand independently and walk at faster speeds. Neuromuscular stimulation (NMS) or electrical stimulation (ES) training is a rehabilitative approach that generates muscle activity, alternating leg extension and flexion even in individuals who are unable to stand or step independently. NMS studies for individuals after SCI have shown improvements in bone density and muscle strength after cycling and resistance training. The main purpose of this study is to address whether stand retraining and NMS compared to stand retraining alone or NMS alone will increase neural and musculoskeletal gains and provide a greater functional recovery towards independent standing.

This project will be completed at two sites: Kessler Foundation Research Center (the grant PI site) and Frazier Rehabilitation Institute, University of Louisville, Kentucky.

DETAILED DESCRIPTION:
There will be three groups in this study. Each group will receive 1.25 hr of intervention per session, for a total of 60 sessions (3 - 4 x week, 15- 20 weeks). Participants in Group 1 will receive 1hr of ES while lying down in the chair followed by 15 min of overground training. Group 2 will receive standing retraining using BWS followed by 15 minutes of overground training. Group 3 will receive standing retraining with ES, followed by 15 min of overground training. Participants will complete the study after 20 weeks of training. The participant will be able to miss 8 consecutive training sessions before being dropped from the study.

PRIMARY AIMS

Specific Aim 1: To examine the effectiveness of standing retraining with ES for alterations in muscle volume (MV) and BMD in the lower limb:

Hypothesis 1.1. SRT with ES compared to SRT alone or ES alone will increase muscle volume(MV) and muscle cross sectional area(MCSA) and potential muscle torque(PMT) at hip, knee and ankle joints (compared to baseline).

Hypothesis 1.2. SRT with ES compared to SRT alone or ES alone will increase absolute BMD in the lower limbs(compared to baseline) Hypothesis 1.3. SRT with ES compared to SRT alone or ES alone will increase markers for bone formation and a decrease in markers for bone resorption commensurate with the observed increase in BMD (compared to baseline) SECONDARY AIMS Specific Aim 2 To examine the effectiveness of standing with ES for improvements in functional outcome and alterations in EMG in lower limb.

Hypothesis 2.1. SRT with ES compared with SRT alone or ES alone will improve functional performance(as measured by standing time on the treadmill and overground) Hypothesis 2.2. SRT with ES compared to SRT alone and ES alone will experience a greater increase in the electromyography (EMG) amplitude for all leg muscles examined (compared to baseline) during standing.

Hypothesis 2.3. LT with ES compared to SRT alone and ES alone will experience significantly greater cardiac output (CO) and/or stroke volume SV (compared to baseline).

.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 58 years old with a neurological SCI level between the C6-T10 level and an impairment grade A, B, or C, according to the American Spinal Injury Association (ASIA) Impairment scale.
* Must have a spinal cord injury that is greater than 6 month or less than 2 years post injury
* Must have score less than 3 on the Modified Ashworth Scale.
* Must be able to tolerate electrical stimulation and must show visible muscle contraction to electrical stimulus
* Must be wheelchair reliant for more than 75% of the time

Exclusion Criteria:

* Bone density measurement (as recorded by the researcher) for knee at or below 0.5755 gm/cm2
* Weigh more than 225 Ibs.
* Taller than 6 feet 3 inches
* Post -menopausal, pregnant or a lactating woman.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2006-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral density | 6 months
  Collected at pre and post

SECONDARY OUTCOMES:
Muscle volume (MRI) | 6 months
  Collected pre and post

CONTACTS AND LOCATIONS:
Overall Officials: Gail Forrest, Ph.D, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided